CLINICAL TRIAL: NCT02413359
Title: Research Study in Patients With COPD in High Risk Population in Japan: Proportion of Overlap Between COPD and Asthma, and the Relationship With COPD Exacerbation
Brief Title: High Risk Populations Among COPD Patients in Japan
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D589BR00033
Record Dates: First submitted 2015-04-07; First posted 2015-04-09 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The patients with complications of COPD and asthma have features mixed with two diseases, COPD and asthma. Therefore, the outcomes are worsened if the patients with COPD have symptoms overlapped with asthma, however, no sufficient data exist in Japan for estimating the prevalence of ACOS in patients with COPD. The primary objective of this NIS is to clarify the proportion of ACOS defined by GINA and GOLD in patients with COPD. The main secondary objectives are To explore the features of history of COPD exacerbations, symptoms, eosinophilic inflammation and patient background in patients with ACOS, to clarify the history of COPD exacerbations in patients with COPD, to evaluate the degrees of eosinophilic inflammation of the respiratory tract in patients with COPD and to evaluate the symptoms in patients with COPD. This is a cross-sectional study targeting COPD patients receiving outpatient treatment and follow-up by physicians in Japan. FSI is scheduled as 2Q 2015 and DBL would be locked by 3Q 2015.

DETAILED DESCRIPTION:
Study Site(s), number of subjects planned Number of study sites planned for this research study (scheduled) 60 (undetermined) Number of subjects planned for this research study (scheduled) 1,100 patients

ELIGIBILITY:
Inclusion criteria

* Patients with a diagnosis of COPD (FEV1/FVC<0.7 confirmed based on the past medical records)
* Patients aged 40 years and over at the diagnosis of COPD
* Outpatient
* 10 or more pack-years of current or former smokers
* Patients who have traceable medical records of COPD (including the results of spirometry) going back more than a year
* Patients who meet any of the following two criteria

  1. Patients who have medical records of the results of spirometry at more than two different time points excluding the time point of COPD exacerbations* for the past 3 years
  2. Patients who can provide the results of reversibility testing for respiratory tract
* Patients who give written informed consent regarding the participation in this study

Exclusion criteria

* Patients currently with COPD exacerbations
* Patients who currently enroll in the other interventional study including clinical trials
* Patients who concurrently develop or have a history of lung cancer
* Patients who are disabled to understand the study procedure or answer the questionnaire (i.e. due to the history of alcohol or drug abuse)

Ages: 40 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of COPD
Sampling Method: Non-Probability Sample
Enrollment: 1016 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Proportion of ACOS defined by The Global Initiative for Asthma (GINA) and The Global Initiative for Chronic Obstructive Lung Disease (GOLD) in patients with COPD receiving outpatient treatment and follow-up by physicians in Japan. | up to 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Atsuhi Yoshida, AstraZeneca, Study Director — Japan - Medical Affairs
Locations (1):
- Takenaka Respiratory Clinic, Takarazuka, Hyōgo, Japan

REFERENCES:
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3712&filename=D589BR00033_redactedCSR.pdf